CLINICAL TRIAL: NCT00712283
Title: A Single Center, Randomized, Double-blind, Placebo-controlled, Parallel Group Design Study to Investigate the Effect of 12,5 mg, 25 mg, 50 mg and 75 mg Neramexane Mesylate IR Tablet on Driving Fitness and Capability to Operate Machines in Healthy Volunteers
Brief Title: Investigate the Effect of Neramexane Mesylate IR Tablet on Driving Fitness and Capability to Operate Machines in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Merz Pharmaceuticals, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: MRZ 92579-0628/1
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: fitness to drive; operate machines; To determine the fitness to drive and operate machines.

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- D (Placebo Comparator): healthy volunteers
  Interventions: Drug: Neramexane mesylate
- C (Active Comparator): healthy volunteers
  Interventions: Drug: Neramexane mesylate
- B (Active Comparator): healthy volunteers
  Interventions: Drug: Neramexane mesylate
- A (Active Comparator): healthy volunteers
  Interventions: Drug: Neramexane mesylate

INTERVENTIONS:
Drug: Neramexane mesylate — tablets Group A: duration: 12,5 mg for 7 days and 25 mg for 8 days Group B: duration: 25 mg for 7 days and 50 mg for 8 days Group C: duration: 50 mg for 7 days and 75 mg for 8 days Group D: duration: placebo for 15 days

SUMMARY:
Determination of the ability to drive and operate machines after single and multiple oral dose of Neramexane as compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers, female and male
* age 21 - 50
* BMI 18 - 30 kg/m2
* experienced drivers with a valid driver's license and at least 3 years of driving practice

Exclusion Criteria:

* any clinically relevant finding on physical examination affecting the study objectives
* clinically relevant abnormalities in the ECG laboratory values
* history or present evidence of clinically relevant metabolic, renal, hepatic, pulmonary or cardiovascular disease, CNS disorders, or disturbance of bleeding diagnosis of malignancy
* females who are pregnant or breastfeeding

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Fitness to drive | 15 days

SECONDARY OUTCOMES:
Psychometric test and motor control tests | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Merz Pharmaceuticals, Frankfurt am Main, Germany